CLINICAL TRIAL: NCT04001205
Title: Effect of Atrial Fibrillation Burden on Long-term Risk of Thromboembolic Complications- the FinCV-4 Study
Brief Title: Atrial Fibrillation Burden and Long-term Risk of Thromboembolic Complications- the FinCV-4 Study
Acronym: FinCV-4
Status: Active, not recruiting | Type: Observational
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Juhani Airaksinen, Professor, Turku University Hospital
Other Study IDs: T75/2019
Record Dates: First submitted 2019-06-21; First posted 2019-06-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Stroke, Ischemic
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke | interventions — Anticoagulation Bridge

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No oral anticoagulation: Patients without oral anticoagulation for AF
- Oral anticoagulation: Patients with long term oral anticoagulation
  Interventions: Drug: Anticoagulation Therapy

INTERVENTIONS:
Drug: Anticoagulation Therapy — Long term oral anticoagulation with VKA (vitamin K antagonist) or NOAC (non-vitamin K oral anticoagulant)
  Groups: Oral anticoagulation

SUMMARY:
This study explores the association of symptomatic episodes of atrial fibrillation (AF) occurrence and long-term risk of thromboembolic complications in a retrospective setting.

DETAILED DESCRIPTION:
The study population consists of the FinCV-dataset, which includes 7660 acute cardioversions for atrial fibrillation. The electronic patient records of FinCV-study patients are reviewed to collect data on anticoagulation, number of cardioversions as well as mortality and stroke data. We seek to explore the possible association between the frequency of AF paroxysms in low stroke risk patients and the occurrence of death, stroke and major bleed as well as the net clinical benefit of anticoagulation. Data collection is performed by reviewing electronic patient records.

ELIGIBILITY:
* primary diagnosis of atrial fibrillation (ICD-10 code I48)
* Cardioversion for acute (<48 h) atrial fibrillation
* >18 years of age
* living within the catchment area of the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Original FinCV study (Airaksinen et al. JACC 2013) eligibility criteria: All patients with a primary diagnosis of atrial fibrillation (ICD-10 code I48) were identified from the institutional discharge registries in the 3 participating hospitals. Emergency clinic admission records and databases were then used to review all patients (>18 years of age) with acute (<48 h) atrial fibrillation who underwent cardioversion during the study period. In addition, only patients living in the hospital catchment area were included to get the adequate follow-up data after the cardioversion.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2025-01-08 (Estimated); Study Completion 2025-01-08 (Estimated)

PRIMARY OUTCOMES:
Death | From the first cardioversion through study completion, an average of 6 years
  Death from any cause
Ischemic stroke or TIA (transient ischemic attack) | From the first cardioversion through study completion, an average of 6 years
  Ischemic stroke or TIA diagnosed by neurologist
Major Bleed | From the first cardioversion through study completion, an average of 6 years
  Major Bleeding complication according to ISTH (International Society on Thrombosis and Haemostasis)

SECONDARY OUTCOMES:
Permanent oral anticoagulation | From the first cardioversion through study completion, an average of 6 years.
  Initiation of permanent oral anticoagulation therapy, information on oral anticoaglation initiation done by reviewing electronic patient records

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Heart Center, Turku, Southwest Finland, Finland

REFERENCES:
- [Background] Airaksinen KE, Gronberg T, Nuotio I, Nikkinen M, Ylitalo A, Biancari F, Hartikainen JE. Thromboembolic complications after cardioversion of acute atrial fibrillation: the FinCV (Finnish CardioVersion) study. J Am Coll Cardiol. 2013 Sep 24;62(13):1187-92. doi: 10.1016/j.jacc.2013.04.089. Epub 2013 Jul 10. PMID 23850908